CLINICAL TRIAL: NCT00047437
Title: Heart Failure: A Controlled Trial Investigating Outcomes of Exercise Training (HF-ACTION)
Brief Title: Exercise Training Program to Improve Clinical Outcomes in Individuals With Congestive Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00017406; U01HL063747 (NIH); U01HL064250 (NIH); U01HL064257 (NIH); U01HL064264 (NIH); U01HL064265 (NIH); U01HL066461 (NIH); U01HL066482 (NIH); U01HL066491 (NIH); U01HL066494 (NIH); U01HL066497 (NIH); U01HL066501 (NIH); U01HL068973 (NIH); U01HL068980 (NIH)
Record Dates: First submitted 2002-10-03; First posted 2002-10-04 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Failure, Congestive
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator)
  Interventions: Behavioral: Supervised Exercise Training Program
- 1 (No Intervention)

INTERVENTIONS:
Behavioral: Supervised Exercise Training Program — Exercise 30 minutes minimum three times per week.
  Arms: 2

SUMMARY:
The purpose of this study is to determine the long-term safety and effectiveness of exercise training for individuals with congestive heart failure (CHF).

DETAILED DESCRIPTION:
BACKGROUND:

CHF affects approximately five million Americans and is the number one cause of hospital admission in individuals over the age of 65. Although exercise training improves several clinical measures in individuals with CHF (e.g., peak VO2, heart rate variability, and plasma norepinephrine levels), it is not known whether exercise training reduces mortality in individuals with CHF.

DESIGN NARRATIVE:

This multicenter randomized study will determine if exercise training reduces mortality and hospitalization rates in individuals with moderate to severe CHF. The secondary objective is to evaluate whether an exercise program designed for individuals with CHF improves quality of life and functioning, is economically advantageous, and prevents medical complications.

Three thousand individuals with moderate to severe CHF will be randomly assigned to either standard medical therapy and education, or standard medical therapy and education plus a supervised exercise training program. The exercise training will include 36 supervised clinic-based training sessions followed by home-based exercise and periodic supervised sessions for reinforcement. Participants assigned to the supervised exercise training program will use either a treadmill or stationary bicycle, which will be provided for them.

Recruitment Status: As of November 9, 2006, HF-ACTION has enrolled 2180 subjects and will conclude enrollment at the end of February, 2007, with an anticipated enrollment of approximately 2300 subjects.

ELIGIBILITY:
Inclusion Criteria:

* LVEF less than or equal to 35%
* New York Heart Association (NYHA) class II, III, or IV CHF diagnosis in the 3 months prior to study entry, with a minimum of 6 weeks of treatment
* Must be on optimal heart failure therapy according to American Heart Association (AHA), American College of Cardiology (ACC), and Heart Failure Society of America (HFSA) heart failure guidelines, including treatment with angiotensin II converting enzyme inhibitors (ACEI) and beta-blocker therapy, or have documentation justifying why optimal therapy is not being used, including intolerance, contraindication, participant preference, or physician's judgment
* Must be on stable doses of medications (e.g., beta-blocker, ACEI, and additional medications as listed in the study guidelines) for 6 weeks prior to study entry
* Must be in stable medical condition and able to begin an exercise program, as determined by study physician

Exclusion Criteria:

* Comorbid disease, behavioral limitations, or other limitations that would interfere with exercise training, or would prevent completion of 1 year of exercise training
* Pregnant or planning to become pregnant in the year following study entry
* Major heart event or heart procedure within the 6 weeks prior to study entry
* Heart procedure or hospitalization for any reason planned in the future
* Expecting to receive a heart transplant in the 6 months following study entry
* CHF caused by significant uncorrected primary valvular disease (except mitral regurgitation secondary to left ventricular dysfunction); if valve replacement has been performed, may not participate for 12 months following the procedure
* CHF caused by congenital heart disease or obstructive cardiomyopathy
* Performance of exercise training at regular intervals (more than once per week) at a moderate to vigorous intensity at any time in the 6 weeks prior to study entry
* Exercise testing results that would prevent safe exercise training, as defined by the American Association of Cardiovascular and Pulmonary Rehabilitation (AACVPR) guidelines, including abnormal blood pressure response, early ischemic changes, and unexpected life-threatening arrhythmia
* Use of fixed-rate pacemakers, pacemakers with inability to attain target heart rates, or automatic implantable cardioverter defibrillator (AICD) devices with heart rate limits set below the target heart rate for exercise training
* Use of an intracardiac device such as an implantable cardioverter defibrillator (ICD) or a cardiac resynchronization therapy pacemaker in the 6 months prior to study entry (must demonstrate stability for 6 weeks post-procedure)
* Primary physician considers placement of an intracardiac device such as an ICD or a cardiac resynchronization therapy pacemaker probable within 6 months of study entry; will be excluded until such device has been placed and 6 weeks of stabilization have passed
* Participation in another clinical trial that may interfere with study participation, follow-up, or data collection, or that may affect cardiovascular morbidity or mortality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2331 (Actual)
Dates: Start 2003-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality and all-cause hospitalization rates (measured at Year 3) | Measured as events occur during the lifespan of the trial.

SECONDARY OUTCOMES:
Changes in peak VO2 | Measured at 3 months, 12 months, and 24 months.
Changes in VE/VCO2 slope | Measured at 3 months, 12 months, and 24 months.
Heart rate at a submaximal work load defined as the end of the exercise test's second stage | Measured at 3 months, 12 months, and 24 months.
Changes in 6-minute walk (measured at Month 3 and Year 1) | Measured at 3 months, 12 months, 24 months, 36 months, and at end of study.
Composite of cardiovascular mortality and cardiovascular hospitalization rates | Measured as events occur during the life of the trial.
Composite of cardiovascular mortality and CHF hospitalization rates | Measured as events occur during the life of the trial.
All-cause mortality rates | Measured as events occur during the life of the trial.
Cardiovascular mortality rates | Measured as events occur during the life of the trial.
All-cause hospitalization rates | Measured as events occur during the life of the trial.
CHF hospitalization rates | Measured as events occur during the life of the trial.
Heart attack rates | Measured as events occur during the life of the trial.
Worsening CHF event rates | Measured as events occur during the life of the trial.
Composite of all-cause mortality, all-cause hospitalization, emergency room visit, and urgent clinic visit for CHF exacerbation rates | Measured as events occur during the life of the trial.
Cost | Measured throughout the life of the trial.
Quality of life | Measured at baseline, months 3, 6, 9, 12, 15, 18, 21, 24, 36, and end of study

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M. O'Connor, Study Chair — Duke University; David J. Whellan, Study Chair — Jefferson Medical College of Thomas Jefferson University
Locations (80):
- United States (65):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Heart Clinic Arkansas, Little Rock, Arkansas
  - Memorial Heart Institute, Long Beach, California
  - Ahmanson-University of California Los Angeles, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - University of California at San Diego Medical Center, San Diego, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Heart and Vascular Clinic of Northern Colorado, Fort Collins, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Veterans Affairs Medical Center, Washington D.C., District of Columbia
  - Southwest Florida Heart Group, Fort Myers, Florida
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Cardiovascular Associates of Augusta, Augusta, Georgia
  - Heart and Lung Group of Savannah, Savannah, Georgia
  - Northwestern University Medical Center, Chicago, Illinois
  - University of Chicago Hospitals, Chicago, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - The Care Group, LLC, Indianapolis, Indiana
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Mid America Heart Institute-Saint Luke's Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Glacier View Cardiology, P.C., Kalispell, Montana
  - Bryan Lincoln General Hospital, Lincoln, Nebraska
  - University of Medicine & Dentistry of New Jersey, New Brunswick, New Jersey
  - Hackensack University Medical Center, Westwood, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Saint Francis Hospital, Roslyn, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Davis Heart and Lung Research Institute, Columbus, Ohio
  - Medical University of Ohio, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Sciences University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Saint Thomas Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Lynchburg General Hospital, Lynchburg, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Madison, Madison, Wisconsin
  - Aurora Health Care, Milwaukee, Wisconsin
- Canada (9):
  - University of Calgary, Calgary, Alberta
  - University of Manitoba Health Sciences Center, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Center, London, Ontario
  - Saint Michaels Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Laval Hospital, Sainte-Foy, Quebec
- France (6):
  - CHU de Caen, Caen
  - Hopital Beaujon Cardiologie, Clichy
  - Hopital Henri Mondor-Service de C, Créteil
  - Hopital Broussais, Paris
  - Centre Cardiologie du Nord, Saint-Denis
  - Hopital Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Whellan DJ, O'Connor CM, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Houston-Miller N, Fleg JL, Schulman KA, Pina IL; HF-ACTION Trial Investigators. Heart failure and a controlled trial investigating outcomes of exercise training (HF-ACTION): design and rationale. Am Heart J. 2007 Feb;153(2):201-11. doi: 10.1016/j.ahj.2006.11.007. PMID 17239677
- [Derived] Hejjaji V, Tang Y, Coles T, Jones PG, Reeve BB, Mentz RJ, Spatz ES, Dunlay SM, Caldwell B, Saha A, Tarver ME, Tran A, Patel KK, Henke D, Pina IL, Spertus JA. Psychometric Evaluation of the Kansas City Cardiomyopathy Questionnaire in Men and Women With Heart Failure. Circ Heart Fail. 2021 Sep;14(9):e008284. doi: 10.1161/CIRCHEARTFAILURE.120.008284. Epub 2021 Sep 1. PMID 34465123
- [Derived] Truby LK, Regan JA, Giamberardino SN, Ilkayeva O, Bain J, Newgard CB, O'Connor CM, Felker GM, Kraus WE, McGarrah RW, Shah SH. Circulating long chain acylcarnitines and outcomes in diabetic heart failure: an HF-ACTION clinical trial substudy. Cardiovasc Diabetol. 2021 Aug 3;20(1):161. doi: 10.1186/s12933-021-01353-z. PMID 34344360
- [Derived] Feng KY, O'Connor CM, Clare R, Alhanti B, Pina IL, Kraus WE, Whellan DJ, Mentz RJ. Greater Pain Severity Is Associated with Worse Outcomes in Patients with Heart Failure. J Cardiovasc Transl Res. 2021 Oct;14(5):984-991. doi: 10.1007/s12265-021-10104-0. Epub 2021 Feb 9. PMID 33564986
- [Derived] Regan JA, Kitzman DW, Leifer ES, Kraus WE, Fleg JL, Forman DE, Whellan DJ, Wojdyla D, Parikh K, O'Connor CM, Mentz RJ. Impact of Age on Comorbidities and Outcomes in Heart Failure With Reduced Ejection Fraction. JACC Heart Fail. 2019 Dec;7(12):1056-1065. doi: 10.1016/j.jchf.2019.09.004. PMID 31779928
- [Derived] Mediano MFF, Leifer ES, Cooper LS, Keteyian SJ, Kraus WE, Mentz RJ, Fleg JL. Influence of Baseline Physical Activity Level on Exercise Training Response and Clinical Outcomes in Heart Failure: The HF-ACTION Trial. JACC Heart Fail. 2018 Dec;6(12):1011-1019. doi: 10.1016/j.jchf.2018.09.012. PMID 30497641
- [Derived] Luo N, O'Connor CM, Cooper LB, Sun JL, Coles A, Reed SD, Whellan DJ, Pina IL, Kraus WE, Mentz RJ. Relationship between changing patient-reported outcomes and subsequent clinical events in patients with chronic heart failure: insights from HF-ACTION. Eur J Heart Fail. 2019 Jan;21(1):63-70. doi: 10.1002/ejhf.1299. Epub 2018 Aug 31. PMID 30168635
- [Derived] Warraich HJ, O'Connor C, Wu A, Coles A, Kraus WE, Pina IL, Whellan DJ, Mentz RJ. Differences Between Patients Enrolled Early and Late During Clinical Trial Recruitment: Insights From the HF-ACTION Trial. Circ Cardiovasc Qual Outcomes. 2018 Jul;11(7):e004643. doi: 10.1161/CIRCOUTCOMES.117.004643. No abstract available. PMID 29980656
- [Derived] Ambrosy AP, Bhatt AS, Stebbins AL, Wruck LM, Fudim M, Greene SJ, Kraus WE, O'Connor CM, Pina IL, Whellan DJ, Mentz RJ. Prevalent digoxin use and subsequent risk of death or hospitalization in ambulatory heart failure patients with a reduced ejection fraction-Findings from the Heart Failure: A Controlled Trial Investigating Outcomes of Exercise Training (HF-ACTION) randomized controlled trial. Am Heart J. 2018 May;199:97-104. doi: 10.1016/j.ahj.2018.02.004. Epub 2018 Feb 11. PMID 29754673
- [Derived] Pokharel Y, Khariton Y, Tang Y, Nassif ME, Chan PS, Arnold SV, Jones PG, Spertus JA. Association of Serial Kansas City Cardiomyopathy Questionnaire Assessments With Death and Hospitalization in Patients With Heart Failure With Preserved and Reduced Ejection Fraction: A Secondary Analysis of 2 Randomized Clinical Trials. JAMA Cardiol. 2017 Dec 1;2(12):1315-1321. doi: 10.1001/jamacardio.2017.3983. PMID 29094152
- [Derived] Sharma A, Stevens SR, Lucas J, Fiuzat M, Adams KF, Whellan DJ, Donahue MP, Kitzman DW, Pina IL, Zannad F, Kraus WE, O'Connor CM, Felker GM. Utility of Growth Differentiation Factor-15, A Marker of Oxidative Stress and Inflammation, in Chronic Heart Failure: Insights From the HF-ACTION Study. JACC Heart Fail. 2017 Oct;5(10):724-734. doi: 10.1016/j.jchf.2017.07.013. PMID 28958347
- [Derived] Ambrosy AP, Cerbin LP, DeVore AD, Greene SJ, Kraus WE, O'Connor CM, Pina IL, Whellan DJ, Wojdyla D, Wu A, Mentz RJ. Aerobic exercise training and general health status in ambulatory heart failure patients with a reduced ejection fraction-Findings from the Heart Failure and A Controlled Trial Investigating Outcomes of Exercise Training (HF-ACTION)trial. Am Heart J. 2017 Apr;186:130-138. doi: 10.1016/j.ahj.2016.12.017. Epub 2017 Jan 19. PMID 28454828
- [Derived] Luo N, Merrill P, Parikh KS, Whellan DJ, Pina IL, Fiuzat M, Kraus WE, Kitzman DW, Keteyian SJ, O'Connor CM, Mentz RJ. Exercise Training in Patients With Chronic Heart Failure and Atrial Fibrillation. J Am Coll Cardiol. 2017 Apr 4;69(13):1683-1691. doi: 10.1016/j.jacc.2017.01.032. PMID 28359513
- [Derived] Kelly JP, Dunning A, Schulte PJ, Fiuzat M, Leifer ES, Fleg JL, Cooper LS, Keteyian SJ, Kitzman DW, Pina IL, Kraus WE, Whellan DJ, O'Connor CM, Mentz RJ. Statins and Exercise Training Response in Heart Failure Patients: Insights From HF-ACTION. JACC Heart Fail. 2016 Aug;4(8):617-24. doi: 10.1016/j.jchf.2016.05.006. Epub 2016 Jul 6. PMID 27395348
- [Derived] Keteyian SJ, Patel M, Kraus WE, Brawner CA, McConnell TR, Pina IL, Leifer ES, Fleg JL, Blackburn G, Fonarow GC, Chase PJ, Piner L, Vest M, O'Connor CM, Ehrman JK, Walsh MN, Ewald G, Bensimhon D, Russell SD; HF-ACTION Investigators. Variables Measured During Cardiopulmonary Exercise Testing as Predictors of Mortality in Chronic Systolic Heart Failure. J Am Coll Cardiol. 2016 Feb 23;67(7):780-9. doi: 10.1016/j.jacc.2015.11.050. PMID 26892413
- [Derived] Ahmad T, Kelly JP, McGarrah RW, Hellkamp AS, Fiuzat M, Testani JM, Wang TS, Verma A, Samsky MD, Donahue MP, Ilkayeva OR, Bowles DE, Patel CB, Milano CA, Rogers JG, Felker GM, O'Connor CM, Shah SH, Kraus WE. Prognostic Implications of Long-Chain Acylcarnitines in Heart Failure and Reversibility With Mechanical Circulatory Support. J Am Coll Cardiol. 2016 Jan 26;67(3):291-9. doi: 10.1016/j.jacc.2015.10.079. PMID 26796394
- [Derived] Cooper LB, Mentz RJ, Sun JL, Schulte PJ, Fleg JL, Cooper LS, Pina IL, Leifer ES, Kraus WE, Whellan DJ, Keteyian SJ, O'Connor CM. Psychosocial Factors, Exercise Adherence, and Outcomes in Heart Failure Patients: Insights From Heart Failure: A Controlled Trial Investigating Outcomes of Exercise Training (HF-ACTION). Circ Heart Fail. 2015 Nov;8(6):1044-51. doi: 10.1161/CIRCHEARTFAILURE.115.002327. PMID 26578668
- [Derived] Fiuzat M, Wojdyla D, Pina I, Adams K, Whellan D, O'Connor CM. Heart Rate or Beta-Blocker Dose? Association With Outcomes in Ambulatory Heart Failure Patients With Systolic Dysfunction: Results From the HF-ACTION Trial. JACC Heart Fail. 2016 Feb;4(2):109-115. doi: 10.1016/j.jchf.2015.09.002. Epub 2015 Oct 28. PMID 26519996
- [Derived] Ahmad T, O'Brien EC, Schulte PJ, Stevens SR, Fiuzat M, Kitzman DW, Adams KF, Kraus WE, Pina IL, Donahue MP, Zannad F, Whellan DJ, O'Connor CM, Felker GM. Evaluation of the Incremental Prognostic Utility of Increasingly Complex Testing in Chronic Heart Failure. Circ Heart Fail. 2015 Jul;8(4):709-16. doi: 10.1161/CIRCHEARTFAILURE.114.001996. Epub 2015 Jun 1. PMID 26034004
- [Derived] Dardas T, Li Y, Reed SD, O'Connor CM, Whellan DJ, Ellis SJ, Schulman KA, Kraus WE, Forman DE, Levy WC. Incremental and independent value of cardiopulmonary exercise test measures and the Seattle Heart Failure Model for prediction of risk in patients with heart failure. J Heart Lung Transplant. 2015 Aug;34(8):1017-23. doi: 10.1016/j.healun.2015.03.017. Epub 2015 Mar 26. PMID 25940075
- [Derived] Mentz RJ, Babyak MA, Bittner V, Fleg JL, Keteyian SJ, Swank AM, Pina IL, Kraus WE, Whellan DJ, O'Connor CM, Blumenthal JA; HF-ACTION Investigators. Prognostic significance of depression in blacks with heart failure: insights from Heart Failure: a Controlled Trial Investigating Outcomes of Exercise Training. Circ Heart Fail. 2015 May;8(3):497-503. doi: 10.1161/CIRCHEARTFAILURE.114.001995. Epub 2015 Apr 21. PMID 25901047
- [Derived] Ahmad T, Pencina MJ, Schulte PJ, O'Brien E, Whellan DJ, Pina IL, Kitzman DW, Lee KL, O'Connor CM, Felker GM. Clinical implications of chronic heart failure phenotypes defined by cluster analysis. J Am Coll Cardiol. 2014 Oct 28;64(17):1765-74. doi: 10.1016/j.jacc.2014.07.979. Epub 2014 Oct 21. PMID 25443696
- [Derived] Jones LW, Douglas PS, Khouri MG, Mackey JR, Wojdyla D, Kraus WE, Whellan DJ, O'Connor CM. Safety and efficacy of aerobic training in patients with cancer who have heart failure: an analysis of the HF-ACTION randomized trial. J Clin Oncol. 2014 Aug 10;32(23):2496-502. doi: 10.1200/JCO.2013.53.5724. Epub 2014 Jul 7. PMID 25002717
- [Derived] Felker GM, Fiuzat M, Thompson V, Shaw LK, Neely ML, Adams KF, Whellan DJ, Donahue MP, Ahmad T, Kitzman DW, Pina IL, Zannad F, Kraus WE, O'Connor CM. Soluble ST2 in ambulatory patients with heart failure: Association with functional capacity and long-term outcomes. Circ Heart Fail. 2013 Nov;6(6):1172-9. doi: 10.1161/CIRCHEARTFAILURE.113.000207. Epub 2013 Oct 8. PMID 24103327
- [Derived] Piccini JP, Hellkamp AS, Whellan DJ, Ellis SJ, Keteyian SJ, Kraus WE, Hernandez AF, Daubert JP, Pina lL, O'Connor CM; HF-ACTION Investigators. Exercise training and implantable cardioverter-defibrillator shocks in patients with heart failure: results from HF-ACTION (Heart Failure and A Controlled Trial Investigating Outcomes of Exercise TraiNing). JACC Heart Fail. 2013 Apr;1(2):142-8. doi: 10.1016/j.jchf.2013.01.005. PMID 23936756
- [Derived] McCullough PA, Barnard D, Clare R, Ellis SJ, Fleg JL, Fonarow GC, Franklin BA, Kilpatrick RD, Kitzman DW, O'Connor CM, Pina IL, Thadani U, Thohan V, Whellan DJ; HF-ACTION Investigators. Anemia and associated clinical outcomes in patients with heart failure due to reduced left ventricular systolic function. Clin Cardiol. 2013 Oct;36(10):611-20. doi: 10.1002/clc.22181. Epub 2013 Aug 8. PMID 23929781
- [Derived] Li Y, Neilson MP, Whellan DJ, Schulman KA, Levy WC, Reed SD. Associations between Seattle Heart Failure Model scores and health utilities: findings from HF-ACTION. J Card Fail. 2013 May;19(5):311-6. doi: 10.1016/j.cardfail.2013.03.008. PMID 23663813
- [Derived] Keteyian SJ, Leifer ES, Houston-Miller N, Kraus WE, Brawner CA, O'Connor CM, Whellan DJ, Cooper LS, Fleg JL, Kitzman DW, Cohen-Solal A, Blumenthal JA, Rendall DS, Pina IL; HF-ACTION Investigators. Relation between volume of exercise and clinical outcomes in patients with heart failure. J Am Coll Cardiol. 2012 Nov 6;60(19):1899-905. doi: 10.1016/j.jacc.2012.08.958. Epub 2012 Oct 10. PMID 23062530
- [Derived] Reed SD, Li Y, Ellis SJ, Isitt JJ, Cheng S, Schulman KA, Whellan DJ. Associations between hemoglobin level, resource use, and medical costs in patients with heart failure: findings from HF-ACTION. J Card Fail. 2012 Oct;18(10):784-91. doi: 10.1016/j.cardfail.2012.08.359. PMID 23040114
- [Derived] Blumenthal JA, Babyak MA, O'Connor C, Keteyian S, Landzberg J, Howlett J, Kraus W, Gottlieb S, Blackburn G, Swank A, Whellan DJ. Effects of exercise training on depressive symptoms in patients with chronic heart failure: the HF-ACTION randomized trial. JAMA. 2012 Aug 1;308(5):465-74. doi: 10.1001/jama.2012.8720. PMID 22851113
- [Derived] Swank AM, Horton J, Fleg JL, Fonarow GC, Keteyian S, Goldberg L, Wolfel G, Handberg EM, Bensimhon D, Illiou MC, Vest M, Ewald G, Blackburn G, Leifer E, Cooper L, Kraus WE; HF-ACTION Investigators. Modest increase in peak VO2 is related to better clinical outcomes in chronic heart failure patients: results from heart failure and a controlled trial to investigate outcomes of exercise training. Circ Heart Fail. 2012 Sep 1;5(5):579-85. doi: 10.1161/CIRCHEARTFAILURE.111.965186. Epub 2012 Jul 6. PMID 22773109
- [Derived] Fiuzat M, Wojdyla D, Kitzman D, Fleg J, Keteyian SJ, Kraus WE, Pina IL, Whellan D, O'Connor CM. Relationship of beta-blocker dose with outcomes in ambulatory heart failure patients with systolic dysfunction: results from the HF-ACTION (Heart Failure: A Controlled Trial Investigating Outcomes of Exercise Training) trial. J Am Coll Cardiol. 2012 Jul 17;60(3):208-15. doi: 10.1016/j.jacc.2012.03.023. Epub 2012 May 2. PMID 22560018
- [Derived] Whellan DJ, Nigam A, Arnold M, Starr AZ, Hill J, Fletcher G, Ellis SJ, Cooper L, Onwuanyi A, Chandler B, Keteyian SJ, Ewald G, Kao A, Gheorghiade M. Benefit of exercise therapy for systolic heart failure in relation to disease severity and etiology-findings from the Heart Failure and A Controlled Trial Investigating Outcomes of Exercise Training study. Am Heart J. 2011 Dec;162(6):1003-10. doi: 10.1016/j.ahj.2011.09.017. PMID 22137073
- [Derived] O'Connor CM, Whellan DJ, Wojdyla D, Leifer E, Clare RM, Ellis SJ, Fine LJ, Fleg JL, Zannad F, Keteyian SJ, Kitzman DW, Kraus WE, Rendall D, Pina IL, Cooper LS, Fiuzat M, Lee KL. Factors related to morbidity and mortality in patients with chronic heart failure with systolic dysfunction: the HF-ACTION predictive risk score model. Circ Heart Fail. 2012 Jan;5(1):63-71. doi: 10.1161/CIRCHEARTFAILURE.111.963462. Epub 2011 Nov 23. PMID 22114101
- [Derived] Felker GM, Fiuzat M, Shaw LK, Clare R, Whellan DJ, Bettari L, Shirolkar SC, Donahue M, Kitzman DW, Zannad F, Pina IL, O'Connor CM. Galectin-3 in ambulatory patients with heart failure: results from the HF-ACTION study. Circ Heart Fail. 2012 Jan;5(1):72-8. doi: 10.1161/CIRCHEARTFAILURE.111.963637. Epub 2011 Oct 20. PMID 22016505
- [Derived] Atchley AE, Iskandrian AE, Bensimhon D, Ellis SJ, Kitzman DW, Shaw LK, Pagnanelli RA, Whellan DJ, Gardin JM, Kao A, Abdul-Nour K, Ewald G, Walsh MN, Kraus WE, O'Connor CM, Borges-Neto S; HF-ACTION Trial Nuclear Ancillary Study Investigators. Relationship of technetium-99m tetrofosmin-gated rest single-photon emission computed tomography myocardial perfusion imaging to death and hospitalization in heart failure patients: results from the nuclear ancillary study of the HF-ACTION trial. Am Heart J. 2011 Jun;161(6):1038-45. doi: 10.1016/j.ahj.2011.02.007. Epub 2011 Apr 6. PMID 21641348
- [Derived] Reed SD, Whellan DJ, Li Y, Friedman JY, Ellis SJ, Pina IL, Settles SJ, Davidson-Ray L, Johnson JL, Cooper LS, O'Connor CM, Schulman KA; HF-ACTION Investigators. Economic evaluation of the HF-ACTION (Heart Failure: A Controlled Trial Investigating Outcomes of Exercise Training) randomized controlled trial: an exercise training study of patients with chronic heart failure. Circ Cardiovasc Qual Outcomes. 2010 Jul;3(4):374-81. doi: 10.1161/CIRCOUTCOMES.109.907287. Epub 2010 Jun 15. PMID 20551371
- [Derived] Keteyian SJ, Isaac D, Thadani U, Roy BA, Bensimhon DR, McKelvie R, Russell SD, Hellkamp AS, Kraus WE; HF-ACTION Investigators. Safety of symptom-limited cardiopulmonary exercise testing in patients with chronic heart failure due to severe left ventricular systolic dysfunction. Am Heart J. 2009 Oct;158(4 Suppl):S72-7. doi: 10.1016/j.ahj.2009.07.014. PMID 19782792
- [Derived] Flynn KE, Lin L, Ellis SJ, Russell SD, Spertus JA, Whellan DJ, Pina IL, Fine LJ, Schulman KA, Weinfurt KP; HF-ACTION Investigators. Outcomes, health policy, and managed care: relationships between patient-reported outcome measures and clinical measures in outpatients with heart failure. Am Heart J. 2009 Oct;158(4 Suppl):S64-71. doi: 10.1016/j.ahj.2009.07.010. PMID 19782791
- [Derived] Atchley AE, Kitzman DW, Whellan DJ, Iskandrian AE, Ellis SJ, Pagnanelli RA, Kao A, Abdul-Nour K, O'Connor CM, Ewald G, Kraus WE, Borges-Neto S; HF-ACTION Investigators. Myocardial perfusion, function, and dyssynchrony in patients with heart failure: baseline results from the single-photon emission computed tomography imaging ancillary study of the Heart Failure and A Controlled Trial Investigating Outcomes of Exercise TraiNing (HF-ACTION) Trial. Am Heart J. 2009 Oct;158(4 Suppl):S53-63. doi: 10.1016/j.ahj.2009.07.009. PMID 19782789
- [Derived] Felker GM, Whellan D, Kraus WE, Clare R, Zannad F, Donahue M, Adams K, McKelvie R, Pina IL, O'Connor CM; HF-ACTION Investigators. N-terminal pro-brain natriuretic peptide and exercise capacity in chronic heart failure: data from the Heart Failure and a Controlled Trial Investigating Outcomes of Exercise Training (HF-ACTION) study. Am Heart J. 2009 Oct;158(4 Suppl):S37-44. doi: 10.1016/j.ahj.2009.07.011. PMID 19782787
- [Derived] Horwich TB, Leifer ES, Brawner CA, Fitz-Gerald MB, Fonarow GC; HF-ACTION Investigators. The relationship between body mass index and cardiopulmonary exercise testing in chronic systolic heart failure. Am Heart J. 2009 Oct;158(4 Suppl):S31-6. doi: 10.1016/j.ahj.2009.07.016. PMID 19782786
- [Derived] Russell SD, Saval MA, Robbins JL, Ellestad MH, Gottlieb SS, Handberg EM, Zhou Y, Chandler B; HF-ACTION Investigators. New York Heart Association functional class predicts exercise parameters in the current era. Am Heart J. 2009 Oct;158(4 Suppl):S24-30. doi: 10.1016/j.ahj.2009.07.017. PMID 19782785
- [Derived] Pina IL, Kokkinos P, Kao A, Bittner V, Saval M, Clare B, Goldberg L, Johnson M, Swank A, Ventura H, Moe G, Fitz-Gerald M, Ellis SJ, Vest M, Cooper L, Whellan D; HF-ACTION Investigators. Baseline differences in the HF-ACTION trial by sex. Am Heart J. 2009 Oct;158(4 Suppl):S16-23. doi: 10.1016/j.ahj.2009.07.012. PMID 19782784
- [Derived] Whellan DJ, Ellis SJ, Kraus WE, Hawthorne K, Pina IL, Keteyian SJ, Kitzman DW, Cooper L, Lee K, O'Connor CM. Method for establishing authorship in a multicenter clinical trial. Ann Intern Med. 2009 Sep 15;151(6):414-20. doi: 10.7326/0003-4819-151-6-200909150-00006. PMID 19755366
- [Derived] Flynn KE, Pina IL, Whellan DJ, Lin L, Blumenthal JA, Ellis SJ, Fine LJ, Howlett JG, Keteyian SJ, Kitzman DW, Kraus WE, Miller NH, Schulman KA, Spertus JA, O'Connor CM, Weinfurt KP; HF-ACTION Investigators. Effects of exercise training on health status in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1451-9. doi: 10.1001/jama.2009.457. PMID 19351942
- [Derived] O'Connor CM, Whellan DJ, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Miller NH, Fleg JL, Schulman KA, McKelvie RS, Zannad F, Pina IL; HF-ACTION Investigators. Efficacy and safety of exercise training in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1439-50. doi: 10.1001/jama.2009.454. PMID 19351941